CLINICAL TRIAL: NCT02739217
Title: A Phase 2, Single-Arm, Open-Label Study to Evaluate the Safety and Tolerability of PBI-4050 and of Its Effects on the Inflammatory, Fibrosis, Diabetes and Obesity Biomarkers in Subjects With Alström Syndrome
Brief Title: Safety and Tolerability of PBI-4050 and Its Effects on the Biomarkers in Subjects With Alström Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI-4050-ATX-9-05
Record Dates: First submitted 2016-02-25; First posted 2016-04-15 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Inflammation and Fibrosis; Diabetes
MeSH Terms: conditions — Inflammation; Fibrosis; Diabetes Mellitus | interventions — setogepram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PBI-4050 (Experimental): Four 200 mg capsules (total 800 mg) administered orally, once daily.
  Interventions: Drug: PBI-4050

INTERVENTIONS:
Drug: PBI-4050 — Four 200 mg capsules (800 mg total) administered orally, once daily.

SUMMARY:
This is a Phase 2, single-centre, single-arm, open-label study of the safety, tolerability, and effects on biomarkers of PBI-4050 in subjects with Alström syndrome for a treatment duration of 24 weeks.

Subjects who complete the initial 24 weeks of treatment may continue treatment for an additional 36 or 48 weeks, provided the subject signs informed consent.

DETAILED DESCRIPTION:
This is a Phase 2, single-centre, single-arm, open-label study of the safety, tolerability, and effects on biomarkers of PBI-4050 in subjects with Alström syndrome. Approximately 18 subjects will be enrolled. The duration of study participation is approximately 35 weeks for each subject and comprises of 9 on site visits and telephone contacts in between visits.

Subjects who complete the initial 24 weeks of treatment may continue treatment for an additional 36 or 48 weeks (Extension Period [EP]), provided the subject signs informed consent. The extension period includes a further 3 on site visits and telephone contacts in between visits. The total duration of the study participation is extended to approximately 71 or 83 weeks. The Data Safety Monitoring Board (DSMB) will determine if the safety data continue to support treatment for an additional 36 or 48 weeks.

At the completion of the EP End of Treatment, subjects will be allowed to enrol in the Alström Rollover Study PBI-4050-CT-9-10 and continue ongoing study medication without any break in treatment.

ELIGIBILITY:
Inclusion Criteria :

* Subject is 16 years of age or older at screening.
* Subject has signed informed consent.
* Subject has a documented diagnosis of Alström syndrome
* Subject on diabetes treatment has been receiving the same antidiabetic agent(s) for a minimum of 1 month before screening.
* Subject is able and willing to self-monitor blood glucose level at home or can obtain adequate assistance from care givers.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening and agree to use adequate birth control from screening throughout the study and for 30 days after the last Investigational Medicinal Product (IMP) administration. If a male subject has not been vasectomized at least 6 months before screening and partners with a woman of childbearing potential, he must be willing to use an acceptable contraceptive method throughout the study and for 30 days after the last IMP administration.

Exclusion Criteria:

* Subject has recent or on-going infection requiring systemic treatment with an anti-infective agent within 30 days before screening.
* Subject has had at least two documented episodes of severe hypoglycaemia within 12 months before screening
* Subject has uncontrolled hypertension with BP > 170/100 mmHg as determined at screening.
* Subject has alanine transaminase (ALT) or aspartate transaminase (AST) level ≥ 5 × upper limit of normal (ULN) at screening.
* Subject is currently using weight loss medications at screening. Subjects may be re-screened after stopping the weight loss medication for a period of at least 5 half-lives.
* Subject has used any moderate/potent inducer or inhibitor of CYP2C9 isozyme or strong inducer or inhibitor of cytochrome P450 (CYP) 3A isozyme within 30 days prior to the first study drug administration.
* Subject has a history of chronic alcohol or other substance abuse as determined at screening.
* Woman who is pregnant, breast-feeding, or planning a pregnancy during the course of the study as determined at screening.
* Subject has any condition that, in the investigator's opinion, is likely to interfere with study conduct and compliance
* Subject has a history of an allergic reaction to PBI-4050 or any of its excipients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Description and number of abnormal laboratory values and adverse events that are related to treatment. | Primary on 24 weeks; Final on all data (including Extension Period)

SECONDARY OUTCOMES:
Change from baseline in metabolic syndrome parameters over time. | 24 weeks and end of Extension Period
  Change from baseline in fasting plasma glucose over time. Change from baseline in fasting plasma insulin over time. Change from baseline in glycated hemoglobin (HbA1c) over time. Change from baseline in Homeostasis Model Assessment for steady state beta cell function (HOMA-B) and insulin sensitivity (HOMA-S) over time.
Change from baseline in biomarkers in blood and urine over time | 24 weeks and end of Extension Phase
  Percentage of reduction and/or increase of level of biomarkers
Change from baseline in cardiac function parameter: NT-proBNP | 24 weeks and end of Extension Phase
Change from baseline of antidiabetic treatment | 24 weeks and end of Extension Phase
  Dosing change, new medication added or treatment discontinuation

OTHER OUTCOMES:
Changes from baseline in histological appearances in fat biopsies | 24 weeks and end of Extension Phase
  Measuring the degree of fibrosis
Changes from baseline in global metabolome and microdialysate fractions | 24 weeks and end of Extension Phase
Change from baseline in the liver stiffness | 24 weeks and end of Extension Phase
  Measured in kilopascal (kPa) correlated to fibrosis by using a FibroScan
Change from baseline in fat content and fibrosis burden in liver MRI | 24 weeks and end of Extension Phase
Change from baseline in left ventricular ejection fraction in cardiac MRI | 24 weeks and end of Extension Phase
Change from baseline in blood glucose as measured by weekly 4 point profile | 24 weeks and end of Extension Phase
Change from baseline in hyperinsulinaemic-euglycaemic clamp measurements. | 24 weeks and end of Extension Phase

CONTACTS AND LOCATIONS:
Overall Officials: Tarekegn Hiwot, MD, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baig S, Veeranna V, Bolton S, Edwards N, Tomlinson JW, Manolopoulos K, Moran J, Steeds RP, Geberhiwot T. Treatment with PBI-4050 in patients with Alstrom syndrome: study protocol for a phase 2, single-Centre, single-arm, open-label trial. BMC Endocr Disord. 2018 Nov 26;18(1):88. doi: 10.1186/s12902-018-0315-6. PMID 30477455